CLINICAL TRIAL: NCT01766375
Title: A Multi-center, Open, Randomized-control Study to Compare the Effects and Safety of Idarubicin-strengthened Pretreatment Program and Conventional Busulfan Cyclophosphamide Pretreatment Program on High-risk Acute Myeloid Leukemia Patient
Brief Title: the Effects and Safety of Idarubicin-strengthened Pretreatment Program and Conventional Busulfan Cyclophosphamide Pretreatment Program on High-risk Acute Myeloid Leukemia Patient
Acronym: IDBUCY
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Lan YongRong, Director of the Hematology department of the First Affiliated Hospital of Guangxi Medical University, Guangxi Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GuangXi-AML- HSCT-2012-07
Record Dates: First submitted 2012-12-28; First posted 2013-01-11 (Estimated); Last update posted 2013-01-11 (Estimated); Status verified 2013-01

CONDITIONS: Acute Myeloid Leukemia
Keywords: idarubicin; busulfan; cyclophosphamide; pretreatment; high-risk acute myeloid leukemia patient
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDBUCY (Experimental): Idarubicin: 20mg/m2 a day, d-12 ~d-10, intravenous infusion for 1 hour. Busulfan: 4mg/Kg a day, oral administration, d-7 ~d-4, or 3.2mg/Kg a day, intravenous infusion, d-7~d-4.
  cyclophosphamide: 60mg/Kg a day, intravenous infusion, d-3~d-2.
  Interventions: Drug: Cyclosporin A,mycophenolate mofetil,Methotrexate
- BUCY (Active Comparator): Busulfan: 4mg/Kg a day, oral administration, d-7 ~d-4, or 3.2mg/Kg a day, intravenous infusion, d-7~d-4.
  Cyclophosphamide: 60mg/Kg a day, intravenous infusion, d-3~d-2.
  Interventions: Drug: Cyclosporin A,mycophenolate mofetil,Methotrexate

INTERVENTIONS:
Drug: Cyclosporin A,mycophenolate mofetil,Methotrexate — GVHD is prevented by CSA+MMF+MTX in sibling allogeneic hematopoietic stem cell transplantation (starting from day -1, 3mg/kg of CSA was infused by continuous intravenous drip until gastrointestinal function returned normal when method of administration was changed to oral administration.

SUMMARY:
This study was a multi-center, open, randomized-control study on the effects and safety of idarubicin 60mg/M2 combined with BUCY pretreatment program or BUCY pretreatment program on the overall survival rate and disease-free survival rate of acute myeloid leukemia patient in high-risk group over a period of 2 years.

DETAILED DESCRIPTION:
This study was a multi-center, open, randomized-control study. It evaluates the effects and safety of idarubicin 60mg/M2 combined with BUCY pretreatment program or BUCY pretreatment program on acute myeloid leukemia patient in high-risk group. 200 patients were studied with 100 patients in each group.

Patients enrolled were randomly divided into group A (idarubicin 60mg/M2 combined with BUCY group) and group B (BUCY group). SAS randomization software was used to obtain randomization numbers. Patients were recommend to start pretreatment within 7 days after randomization.

Main objective: 2-year overall survival (OS) and disease-free survival (DFS) rates.

Secondary objective: safety evaluation (early complications of transplantation, liver, kidney and heart toxicity, treatment-related mortality, blood recovery time), the median period of disease-free survival.

Test drugs Idarubicin (Zavedos ®, Pfizer), busulfan, cyclophosphamide.

Pretreatment plan Drug Group A (IDA 60mg/M2 + BUCY) Group B (BUCY) IDA: 20mg/m2 a day, d-12 ~d-10, intravenous infusion for 1 hour. BU: 4mg/Kg a day, oral administration, d-7 ~d-4, or 3.2mg/Kg a day, intravenous infusion, d-7~d-4.

CY: 60mg/Kg a day, intravenous infusion, d-3~d-2. GVHD prevention plan GVHD is prevented by CSA+MMF+MTX in sibling allogeneic hematopoietic stem cell transplantation (starting from day -1, 3mg/kg of CSA was infused by continuous intravenous drip until gastrointestinal function returned normal when method of administration was changed to oral administration. 5mg/kg was divided into twice oral intakes, maintaining cyclosporine concentration at 200-300ug / L; MTX 15mg/m2 at day +1, 10mg/m2 at day +3, +6 and day +11 (based on actual situations day 11 can be omitted); MMF 0.25g BID starting from day 0 and continued for a month ). Unrelated allogeneic hematopoietic stem cell transplantation used CSA MMF MTX ATG for the prevention of GVHD. 3mg/kg CSA was infused through continuous intravenous drip since day -1 until gastrointestinal function returned to normal when the administration method was changed to oral. 5mg/kg was divided to twice oral intakes maintaining cyclosporine concentrations at 200-300ug/L; MTX 15mg/m2, at day +1, 10mg/m2 at day +3, day +6 and day +11 (based on actual situations day 11 can be omitted); MMF 0.5g BID starting from day 0 and continued for 3 months (a month later, dose can be reduced according to the hemogram); the total ATG was 6mg/kg and was taken in three days, from day -4 to day -2.

Relapse intervention Routine preventive DLI is not recommended, however, if tendency of recurrence found during monitor, chemotherapy, immunotherapy, targeted therapy, secondary transplantation, etc. can be used, and intervention treatment start time should be recorded as the end time.

The efficacy evaluation time point

1. 1-3, 6, 12, 18, 24 months after transplantation.
2. Follow-up evaluation: indicators such as blood routines and bone marrow detection, and minimal residual disease detection after the end of treatment should be done regularly.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18～50;
2. Received peripheral blood hematopoietic stem cell transplantation from siblings or unrelated allogeneic donors with identical matching of HLA or 1 alleles mismatched.
3. Diagnosis: refer to 2011 edition of AML China Guideline for the diagnosis and treatment and diagnosis standards of high-risk acute myeloid leukemia developed through literatures (see Appendix B);
4. Under general condition, ECOG score ≤ 1;
5. Normal cardiac functions;
6. Normal liver and renal function: blood bilirubin≤35 μ mol\/L, AST/ALT lower than twice in the upper limit of normal value, serum creatinine≤ 150 μ mol\/L;
7. Subjects have signed the informed consent form.

Exclusion Criteria:

1. Severe uncontrolled infection before transplantation;
2. With contraindications of idarubicin;
3. Reached the maximum cumulative dose of anthracyclines, for instance, DNR≥ 450mg/m2, mitoxantrone≥140mg/m2, the total cumulative dose of idarubicin≥ 300mg/m2;
4. The other conditions that do not meet the inclusion criteria.

Withdrawal criteria:

1. Those do not meet the inclusion criteria or meet the exclusion criteria after reviewing;
2. Patient withdraws the informed consent form;
3. Patient violates the clinical study protocol;
4. Patient experiences severe adverse events that treatment has to be terminated;
5. Patient that considered no longer fit to complete clinical trials by researchers.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-08; Primary Completion 2016-01 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
2-year disease-free survival (DFS) rates | 4 years
  The purpose of this study is to evaluates the effects of idarubicin 60mg/M2 combined with BUCY pretreatment program or BUCY pretreatment program on acute myeloid leukemia patient in high-risk group.

SECONDARY OUTCOMES:
2-year overall survival (OS) rates | 4 years
  It evaluates the effects of idarubicin 60mg/M2 combined with BUCY pretreatment program or BUCY pretreatment program on acute myeloid leukemia patient in high-risk group. 200 patients were studied with 100 patients in each group

OTHER OUTCOMES:
safety of idarubicin 60mg/M2 combined with BUCY pretreatment program or BUCY pretreatment program | 4 years
  safety evaluation (early complications of transplantation, liver, kidney and heart toxicity, treatment-related mortality, blood recovery time),

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi, China